CLINICAL TRIAL: NCT00165256
Title: Wide Excision Alone for DCIS-Grades 1 and 2
Brief Title: Wide Excision Alone as Treatment for Ductal Carcinoma in Situ of The Breast
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Julia S. Wong, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 94-151
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ductal Carcinoma in Situ of the Breast
Keywords: Ductal carcinoma in situ; DCIS; wide excision
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observation (omission of RT) (Experimental): Wide excision of DCIS; no radiotherapy (RT).
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Wide excision of DCIS and a minimum of 1cm histologically negative margin of breast tissue

SUMMARY:
The purpose of this study is to determine if wide excision (surgical removal) alone is adequate treatment for small, grade 1 or 2 ductal carcinoma in situ (DCIS) of the breast.

DETAILED DESCRIPTION:
* Patients with DCIS are usually treated with the combination of breast-conserving surgery and radiation therapy or breast-conserving surgery alone. The purpose of this study is to evaluate whether localized low- or intermediate-grade DCIS, diagnosed with modern mammography and careful pathologic evaluation, could be treated with wide excision alone (omission of radiation therapy) and result in acceptably low local recurrence rates.
* Follow-up consists of physical examinations at least every 6 months by the surgeon or radiation oncologist. Mammograms of the affected breast will be obtained every 6 months for 5 years and then annually. Mammograms of the unaffected breast will be performed annually.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have high quality mammogram including magnification views of the area containing suspicious calcifications.
* A specimen radiograph is required. If the specimen radiograph does not assure removal of all suspicious microcalcifications, a post-operative mammogram showing removal of all suspicious calcifications is required.
* The clinical extent of DCIS must be less than or equal to 2.5 cm.
* Grade 1 or 2 DCIS; patients with lobular carcinoma-in-situ (LCIS) in addition to DCIS in the breast are eligible. Negative margins are not required on the LCIS.
* Patients must undergo a wide excision. A re-excision after the initial biopsy might be needed. Complete resection of the area of DCIS with a histologic margin of at least 1 cm must be achieved.
* Patients must be enrolled on this protocol within 3 months of the last surgical procedure.

Exclusion Criteria:

* Patients with invasive carcinoma including microinvasive disease
* Carcinoma found in the sampled lymph nodes if axillary dissection is done
* Patients with nipple discharge
* Patients with adjuvant chemotherapy or Tamoxifen
* Patients with a history of prior malignancies other than squamous or basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Patients with a history of ipsilateral or contralateral breast carcinoma or DCIS or simultaneous bilateral DCIS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 1995-05; Primary Completion 2002-07 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To determine if patients with DCIS can be effectively treated with wide excision alone. | TBD-survivorship
  Using information gathered from follow-up physical examinations and mammography to check for recurrence (DCIS or invasive carcinoma in the breast), DCIS patients treated with wide excision alone will be evaluated.

SECONDARY OUTCOMES:
To explore whether patients with grade 2 DCIS have a higher breast recurrence than patients with grade 1 DCIS. | TBD-survivorship
  Using information gathered from follow-up physical examinations and mammography, the exploration of breast recurrences between grade 2 DCIS and grade 1 DCIS patients will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wong, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong JS, Kaelin CM, Troyan SL, Gadd MA, Gelman R, Lester SC, Schnitt SJ, Sgroi DC, Silver BJ, Harris JR, Smith BL. Prospective study of wide excision alone for ductal carcinoma in situ of the breast. J Clin Oncol. 2006 Mar 1;24(7):1031-6. doi: 10.1200/JCO.2005.02.9975. Epub 2006 Feb 6. PMID 16461781
- [Result] Wong JS, Chen YH, Gadd MA, Gelman R, Lester SC, Schnitt SJ, Sgroi DC, Silver BJ, Smith BL, Troyan SL, Harris JR. Eight-year update of a prospective study of wide excision alone for small low- or intermediate-grade ductal carcinoma in situ (DCIS). Breast Cancer Res Treat. 2014 Jan;143(2):343-50. doi: 10.1007/s10549-013-2813-6. Epub 2013 Dec 18. PMID 24346130